CLINICAL TRIAL: NCT07117578
Title: Assessment of Preoperative Anxiety in Adult Patient Undergoing Elective Surgery in Eastem Sub-urban Area ofNepa
Brief Title: Preoperative Anxiety in Eastern Nepal (PAEN)
Acronym: PAEN
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Sujan Dhakal, MD, Consultant Anesthesiologist, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: NHRC-562/2024; 562/2024 (Other: Nepal Health Research Council)
Record Dates: First submitted 2025-08-03; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Preoperative Anxiety; Elective Surgery; Clinician Attention
Keywords: APAIS; Clinician Rated Score; Clinician reported anxiety; Elective Surgery; Preoperative Anxiety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Elective Surgery Patients: Adult Elective Surgery Patients in Eastern Suburban Nepal presenting for elective surgery after preoperative anaesthetic checkup and clearance and perioperative counseling.

SUMMARY:
This study is looking at how many adults feel nervous or worried before planned surgery at two hospitals in eastern Nepal. We will include men and women aged 18 to 80 who are having elective operations.

On the day of the preoperative check, the participant will be asked to complete a very short, six-question survey about how anxious the participant feels and how much information the participant wants. It takes about five minutes, and the participant can answer by choosing responses like "not at all," "somewhat," or "extremely."

The investigating anesthesiologist will also make a quick, private note of how anxious they think you are based on their routine pre-anaesthesia check. All of the participant answers and the doctor's note will be kept strictly confidential and stored securely.

Joining the study is entirely voluntary. Deciding not to take part or choosing to leave the study at any time will not change the medical care you receive. There are no extra costs or medical tests beyond what you would normally have.

By sharing your experience, the participant helps us understand what makes patients feel anxious before surgery and how the investigators can improve support and information for future patients.

DETAILED DESCRIPTION:
This is a cross-sectional observational study conducted at Bhadrapur Provincial Hospital and Om Sai Pathibhara Hospital. We aim to enrol 422 adult patients (18-80 years old) with ASA physical status I to III scheduled for elective surgery.

The investigator will use the Amsterdam Preoperative Anxiety and Information Scale (APAIS) to measure patient-reported anxiety and information need. This six-item tool yields an anxiety score (4-20 points) and an information-need score (2-10 points). A score of 11 or more indicates high anxiety. In addition, the attending anesthesiologist will rate each patient's anxiety immediately after the pre-anaesthetic check.

We will collect demographic and clinical data, including age, gender, marital status, education level, occupation, previous anaesthesia exposure, type of anaesthesia, and area of residence. Data entry will be done in Excel, and analysis will be carried out using SPSS. We will report median and interquartile ranges for APAIS scores and use multivariable logistic regression to identify factors associated with high anxiety.

The study protocol has been approved by the Nepal Health Research Council. Participant confidentiality will be maintained through coded identifiers, locked physical records, and encrypted digital files.

The investigator's goal is to determine how common preoperative anxiety is and which patient characteristics influence it. The findings will guide the development of targeted interventions and information programmes to reduce anxiety before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years
* Scheduled for elective surgery with prior pre-anesthetic clearance
* Able to provide informed consent

Exclusion Criteria:

* Decline to participate
* Documented psychiatric disorders or cognitive impairment
* Current treatment with anxiolytics or antidepressants
* Language barrier preventing questionnaire completion
* ASA Physical Status IV or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will involve adult patients (18 years and older) scheduled for elective surgical procedures under general, regional, or combined anesthesia at Bhadrapur Provincial Hospital and Om Sai Pathibhara Hospital in Eastern Suburban Nepal. Recruitment will occur over four months using consecutive sampling. Eligible patients must be classified as American Society of Anesthesiologists (ASA) physical status I-III, able to communicate in Nepali or English, and willing to provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Preoperative Anxiety Prevalence | Single preoperative assessment before surgery
  Assessment Tool: Amsterdam Preoperative Anxiety and Information Scale (APAIS) to measure patient-reported anxiety and information need. This six-item tool yields an anxiety score (4-20 points) and an information-need score (2-10 points).
  Definition: Amsterdam Preoperative Anxiety and Information Scale, total anxiety score ≥11,

SECONDARY OUTCOMES:
Clinician Anxiety Rating Score vs. Amsterdam Preoperative Anxiety and Information Scale | Single preoperative assessment before surgery
  Comparison of the anesthesiologist's subjective rating (CRS), which is a similar scale to APAIS to measure anxiety and information need by the anesthesiologist according to the patient's answer and other objective variables from attached monitors. This six-item tool yields an anxiety score (4-20 points) and an information-need score (2-10 points).
Anxiety Associations with Demographic & Clinical Factors | Single preoperative assessment before Surgery
  Variables: Age, gender, marital status, occupation, education, ASA PS, prior surgery/anesthesia, anesthesia type, region of residence
  Statistical Analysis: Logistic regression

CONTACTS AND LOCATIONS:
Locations (1):
- Om Sai Pathibhara Hospital and Provincial hospital Bhadrapur, Bhadrapur, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No